CLINICAL TRIAL: NCT01632020
Title: Pilot Study: Effect of Metformin on Biomarkers of Colorectal Tumor Cell Growth
Brief Title: Effect of Metformin on Biomarkers of Colorectal Tumor Cell Growth
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 134190
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal tumor; colorectal cancer; colorectal carcinoma; neoplasms, colorectal; Metformin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 2 capsules by mouth twice daily; minimum of 10 days, maximum of 21 days
  Interventions: Drug: Placebo
- Metformin (Active Comparator): Metformin 850 mg (2 capsules) by mouth twice daily; minimum of 10 days, maximum of 21 days
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo — 2 capsules by mouth twice daily; minimum of 10 days, maximum of 21 days
  Other Names: inactive drug
  Arms: Placebo
Drug: Metformin — 850 mg (2 capsules) by mouth twice daily; minimum of 10 days, maximum of 21 days
  Other Names: Glucophage; Glucophage XR; Glumetza; Fortamet; Riomet
  Arms: Metformin

SUMMARY:
The purpose of this study is to investigate the effects of short term oral Metformin therapy on biomarkers for tumor growth in subjects with newly diagnosed colon or rectal adenocarcinoma.

It is hypothesized that there are independent actions of Metformin on the outcome of subjects with colorectal cancer (CRC). Also hypothesized is that metformin effects on CRC cell growth will correlate with this drug's effects on markers mentioned above, because the markers are closely related to tumor growth and metastases.

DETAILED DESCRIPTION:
This is a randomized, double-blinded placebo controlled clinical investigation of the effects of short term oral Metformin therapy on biomarkers for tumor growth in subjects with newly diagnosed colon or rectal adenocarcinoma. Metformin is a well-tolerated drug widely prescribed for treatment of Type 2 diabetes mellitus. Preliminary studies have generated the hypothesis that metformin may have positive effects on both prevention and survival of colon cancer subjects. Clinical trials are ongoing to explore this possibility in breast cancer (NCT01101438). This investigation is the first study of Metformin in colorectal cancer (CRC) patients, and is designed to understand the mechanism of its anti-cancer actions, if any, and its interactions with biomarkers in colorectal cancer patients.

Based upon epidemiological studies, it is hypothesized that there are independent actions of Metformin on the outcome of subjects with CRC. Also hypothesized is that metformin effects on CRC cell growth will correlate with this drug's effects on markers mentioned above, because the markers are closely related to tumor growth and metastases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, all races and ethnicities are eligible
* Age equal to or greater than 18 years of age
* All subjects should have a pathological/histological diagnosis of colorectal cancer.
* Clinical diagnosis of stage I, II, III or IV colon cancer or stage I, II, III or IV rectal cancer; cancer may be primary including a secondary primary
* Candidate for elective surgery(for removal of primary) or endoscopic biopsy
* ECOG Performance status of 0 - 2
* Adequate renal, liver, and bone marrow function
* Hb: (adequate for surgical intervention, with transfusion if necessary)
* WBC: (normal range)
* Platelets: (180K/cmm)
* LFTs: Normal bilirubin (< 2.0mg/dL), AST/ALT (2xULN)
* Renal function: normal creatinine
* Subjects must have signed informed consent
* Female subjects must either not be of child-bearing potential or must have a negative urine pregnancy test within 7 days of beginning the drug or placebo treatment. Subjects are considered not of child-bearing potential if they are surgically sterile or they are postmenopausal for greater than 12 months.

Exclusion Criteria:

* Previously diagnosed with diabetes mellitus Type 1 or Type 2.
* Currently taking biguanides, sulfonylurea drugs, thiazolidinediones, insulin, or mTOR inhibitors or having taken any of these medications during the 12 weeks prior to study participation.
* Currently taking any non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin and unable to stop such medications due to a present medical condition.
* Clinical symptoms of gastrointestinal obstruction or bleeding and consideration for immediate surgery or immediate neoadjuvant chemoradiation.
* Familial Adenomatous Polyposis (FAP), hereditary non-polyposis colorectal cancer (HNPCC), Putz-Jeghers disease, ulcerative colitis, or Crohn's disease.
* Pregnant or lactating.
* History of lactic or other metabolic acidosis.
* Known hypersensitivity to Metformin.
* Uncontrolled infectious disease.
* History of Positivity for human immunodeficiency virus (HIV).
* History of congestive heart failure requiring pharmacologic treatment.
* History of excessive alcohol abuse, defined by a habitual intake of more than three drinks daily.
* Previous or concurrent malignancies, except non-melanoma skin cancers, unless curatively treated and with no evidence of recurrence for > 5 years, with the exception of prior CRC which has been treated and the patient has been in remission and the current primary tumor is a second CRC.
* Unable to swallow and retain oral medication.
* Mal-absorption syndrome, disease affecting gastrointestinal function, or previous resection of the stomach or small bowel.
* Current use of medications for weight loss.
* Currently taking cimetidine, thiazide diuretics or cephalexin. If a patient needs some of these agents, alternative agents should be substituted.
* If the physician feels that the candidate is not suitable for the study, he/she will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rangaswamy Govindarajan, MD, Principal Investigator — University of Arkansas; Frank Simmen, PhD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - Central Arkansas Veterans Heathcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open for enrollment between 7/13/2012 and 3/5/2014. Subjects were recruited from medical clinics at the University of Arkansas for Medical Sciences (UAMS) and the Central Arkansas Veterans Healthcare System (CAVHS).
Pre-assignment Details: There were no significant events following participant enrollment, prior to group assignment.
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 4 | 3
Completed | 2 | 3
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 57 [52 to 61] | 44 [37 to 54] | 49 [37 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proliferation Status of CRC Tumor and Adjacent Normal Tissue Following Metformin Therapy
Time Frame: 10-21 days
Population: Data not collected due to inadequate subject accrual. Analysis not completed.
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Mucosal Apoptotic Status of CRC Tumor and Adjacent Normal Tissue Following Metformin Therapy
Time Frame: 10-21 days
Population: Data not collected due to inadequate subject accrual. Analysis not completed.
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Metformin (N=3)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdomen Pain Not Otherwise Specified (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain of the extremities/ limbs (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects. Outcome measures not computed because data would not be statistically relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes